CLINICAL TRIAL: NCT05677581
Title: Longitudinal Study on the Influence of Iodine Nutrition Status on Thyroid Function of Childbearing Age Women During Pregnancy and 6 Weeks Postpartum
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SF2022-2-2029
Record Dates: First submitted 2022-11-30; First posted 2023-01-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2023-11

CONDITIONS: Thyroid Function; Iodine Nutrition Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pregnancy and lactation period women
  Interventions: Other: iodine nutrition status
- healthy women of childbearing age
  Interventions: Other: iodine nutrition status

INTERVENTIONS:
Other: iodine nutrition status — iodine nutrition status

SUMMARY:
The goal of this observational study is to provide a reference for formulating individual appropriate iodine intake programs for women during pregnancy and postpartum and improving the monitoring and evaluation system of maternal iodine nutrition status. The main questions it aims to answer are:

* To analyse the longitudinal changes of urinary iodine, urinary iodine/creatinine ratio, thyroid function and related factors in different periods of early, middle, late pregnancy and 6 weeks postpartum in Beijing area.
* To explore the relationship between iodine nutrition status and the changes of thyroid function and to further clarify the effect of iodine nutrition status on thyroid function of women of childbearing age during pregnancy and postpartum in combination with dietary intake of iodine questionnaire.

Participants will be detected there thyroid function, the level of median urinary iodine and urinary iodine/creatinine.

Researchers will compare healthy women of childbearing age served as the control group in the same period.

ELIGIBILITY:
8-12 weeks healthy maternal:

Inclusion Criteria:

* primigravida
* no chronic hypertension, thromboembolic disease, severe gastrointestinal, cardiopulmonary and liver diseases before pregnancy
* no systemic lupus erythematosus, rheumatic diseases and other connective tissue diseases or immune diseases before pregnancy
* no adrenocortical hyperplasia, pituitary endocrine diseases and other diseases before pregnancy

Exclusion Criteria:

* multiple pregnancies and multigravida
* a history of type I or type II diabetes before pregnancy
* a clear history of thyroid diseases before pregnancy
* taking drugs that affect thyroid function and/or blood sugar before or during early pregnancy

Healthy women of childbearing age:

Inclusion Criteria:

* 20-40 years old
* no chronic hypertension, thromboembolic disease, severe gastrointestinal, cardiopulmonary and liver diseases
* no systemic lupus erythematosus, rheumatic diseases and other connective tissue diseases or immune diseases
* no adrenocortical hyperplasia, pituitary endocrine diseases and other diseases

Exclusion Criteria:

* a history of type I or type II diabetes
* a clear history of thyroid diseases
* taking drugs that affect thyroid function and/or blood sugar

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: maternal and women of childbearing age in Beijing area
Sampling Method: Non-Probability Sample
Enrollment: 2100 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Data of pregnant women in the early trimester of pregnancy | Any day between weeks 8 and 12 of gestation
  detect the level of serum TSH, FT4, TPOAb, TGAb and the level of median urinary iodine and urinary iodine/creatinine
Data of pregnant women in the middle trimester of pregnancy | Any day between weeks 24 and 28 of gestation
  detect the level of serum TSH, FT4, TPOAb, TGAb and the level of median urinary
Data of pregnant women in the third trimester of pregnancy | Any day between weeks 36 of gestation to the day before parturition
  detect the level of serum TSH, FT4, TPOAb, TGAb and the level of median urinary
Data of postpartum women | 6 weeks after parturition
  detect the level of serum TSH, FT4, TPOAb, TGAb and the level of median urinary

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital ,Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No